CLINICAL TRIAL: NCT03160729
Title: High vs Low Dose Dexamethasone on Complications in the Immediate Postoperative Phase After Nephrectomy (DEX-NEF)
Brief Title: High vs Low Dose Dexamethasone on Complications in the Immediate Postoperative Phase After Nephrectomy
Acronym: DEX-NEF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment, schanges in standard treatment
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristin Julia Steinthorsdottir, MD, clinical assistant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEXNEF01
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Kidney Diseases; Postoperative Complications
MeSH Terms: conditions — Kidney Diseases; Postoperative Complications | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose (Active Comparator): Dexamethasone 24 mg
  Interventions: Drug: Dexamethasone
- Low dose (Active Comparator): Dexamethasone 8 mg
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — pre-operative, single-shot injection

SUMMARY:
The aim of this study is to investigate the effect of a single preoperative high-dose steroid injection on complications in the immediate postoperative phase after open kidney surgery (kidney resection, heminephrectomy, nephrectomy). Primary outcome is complications in the post anaesthesia care unit (PACU). Secondary outcomes are organospecific complications in the post anaesthesia phase, pain and nausea the first 5 days, seroma and wound infection the first 14 days and readmissions the first 30 days after surgery.

The investigators hypothesize that the frequency of transfer to the PACU and organospecific complications will be lower among patients receiving high dose dexamethasone. The investigators hypothesize, that there will be no difference in wound infections, seroma or readmissions.

DETAILED DESCRIPTION:
Post-surgery, patients are traditionally observed and treated in post-anesthesia care units (PACU) until they are discharged to the ward (or directly home) assessed by standardized international discharge criteria.

The research project "Why in PACU?" (Rigshospitalet, Denmark), has since the beginning of 2016 systematically collected and analyzed procedure-related complications in the recovery phase. The complications include pain, nausea/vomiting, circulatory and respiratory problems, orthostatic intolerance and cognitive disorders. Common to all the above-mentioned post-operative problems are the possible links to the inflammatory response caused by the surgical trauma.

Glucocorticoids can in this context be central for the reduction of acute postoperative organ dysfunctions, caused by the anti-inflammatory effect. In a number of different surgical procedures, single dose, pre-operative glucocorticoids have been shown to reduce post-operative nausea and vomiting (PONV), acute pain and need of opioids as well as accelerate the convalescence.

Meta-analyses also showed that single-dose administration of glucocorticoids (methylprednisolone and dexamethasone) for surgical patients is safe as opposed to long-term treatment.

The "Why in PACU?" database shows that 60 % of patients having open kidney surgery have complications in the PACU (primarily pain and hypoxia).

Based on positive results in other procedure-specific studies, all donor-nephrectomy patients at Rigshospitalet, have received pre-operative high-dose steroids, in the form of 24 mg dexamethasone injection since mid-2015. This has resulted in a reduction of pain requiring treatment with 30 %.

Prior to creating clinical recommendations and standards, it is required that the results be tested in a randomized, controlled, clinical trial.

The study is not placebo-controlled since the positive effects of dexamethasone 8 mg on PONV have been shown in numerous trials, and is already being administered to all patients at the clinic. It would therefore not be ethically correct to withdraw from this practise

ELIGIBILITY:
Inclusion Criteria:

Planned open kidney resection, heminephrectomy, nephrectomy Signed informed consent

Exclusion Criteria:

* chronic/ongoing use of glucocorticoids (except inhalation therapy)
* ongoing use of immunosuppressive therapy
* insulin dependent diabetes
* pregnancy/breastfeeding
* allergies toward study medication, or medication in a standard treatment
* previous kidney resection on same side
* thrombectomy in vena cava above diaphragma
* surgery cannot be performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Post-operative complications | 24 hours
  Complications requiring treatment in the PACU

SECONDARY OUTCOMES:
Length of stay, PACU | 24 hours
  Total length of stay in PACU
Length of stay, hospital | 1 month
  Total length of stay in hospital
Discharge score | 1 hour
  Discharge score (according to discharge criteria) in the operating theater
Discharge score | 24 hours
  Discharge score (according to discharge criteria) in the PACU
Complications | 24 hours
  Complications requiring treatment in the ward
Pain postoperative | 4 days
  Self-reported pain (worst and average, days 0-4). Questionnaire.
Analgesics | 4 days
  Self-reported use of pain medication other than standard treatment (days 0-4). Questionnaire.
Post operative nausea and vomiting (PONV) | 4 days
  Self-reported ponv (worst and average, days 0-4. Questionnaire.
Antiemetics | 4 days
  Use of antiemetics other than standard treatment (days 0-4. Questionnaire.
Sleep | 4 days
  Self-reported quality of sleep (days 0-4). Questionnaire.
Mental status | 4 days
  Self-reported feelings of anxiety, unrest, sadness (days 0-4). Questionnaire.
Wound complications | 30 days
  Wound complications/infections
Readmissions | 30 days
  Any readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Kristin J Steinthorsdottir, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No